CLINICAL TRIAL: NCT07273123
Title: Effect of Sugar-Free Chewing Gum Mastication on Fatigue of the Masticatory Muscles in Young Adults With and Without Temporomandibular Joint Disorders
Brief Title: The Effect of Prolonged Sugar-Free Chewing Gum Mastication on Self-Reported Fatigue Levels and Changes of Static and Dynamic Surface Electromyography Parameters in Young Individuals With and Without Temporomandibular Joint Disorders.
Status: Recruiting | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Aesha Allam, DDS, University of Milan
Other Study IDs: 95 /25
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Temporomandibular Joint Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Case group (subjects with TMD): This group contains subjects with temporomandibular disorders
  Interventions: Other: Mastication of sugar-free chewing gum
- Control group (TMD-free subjects): This group contains healthy subjects without temporomandibular disorders
  Interventions: Other: Mastication of sugar-free chewing gum

INTERVENTIONS:
Other: Mastication of sugar-free chewing gum — The chewing task will last for a maximum of 18 minutes.

SUMMARY:
This case-control study investigates fatigue induced by prolonged gum mastication in individuals with temporomandibular disorders (TMD). The study addresses two primary questions:

How does self-reported fatigue, measured with a visual analogue scale (VAS), change during sustained chewing? How do static and dynamic surface electromyographic (sEMG) parameters evolve over the same period? Participants with TMD will be compared with healthy controls to determine group differences in perceived fatigue and EMG responses.

All participants will undergo baseline EMG assessment, then chew sugar-free gum continuously for 3 minutes, alternating sides without rest. After each 3-minute interval, static and dynamic EMG recordings will be obtained and participants will rate their fatigue on the VAS. This cycle may be repeated up to six times (maximum 18 minutes). Participants are free to stop chewing at any time if fatigue becomes intolerable.

ELIGIBILITY:
Inclusion criteria (both groups):

* Age 19-35 years
* Chewing-gum users, even occasional
* Good general health
* Good oral health

Inclusion criteria (Healthy controls):

- no diagnosed temporomandibular joint disorders

Inclusion criteria (study group)

- diagnosed temporomandibular joint disorders

Exclusion criteria (both groups):

* Non chewing gum users
* History of neurological disorders
* History of musculoskeletal diseases
* History of facial or cervical injuries
* Presence of cervical pain
* Two or more missing teeth
* Current treatment with fixed or removable orthodontic appliances
* Active periodontal disease
* Presence of cavitated carious lesions

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of volunteer participants recruited from the undergraduate dentistry program and postgraduate specialty training programs at the University of Milan.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported (subjective) fatigue after prolonged sugar-free chewing gum mastication | 18 minutes

SECONDARY OUTCOMES:
Changes of static and dynamic surface electromyography (sEMG) parameters after prolonged mastication of sugar-free chewing gum | 18 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milan, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes